CLINICAL TRIAL: NCT02946021
Title: Assessment of Lymphatic Structure and Function Pre- and Post- Treatment and During Recovery in Head and Neck Cancer Patients Using NIR Fluorescence Lymphatic Imaging
Brief Title: Response to Intermittent Pneumatic Compression Therapy in Head and Neck Cancer-Related Lymphedema
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tactile Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-16-0465
Record Dates: First submitted 2016-10-20; First posted 2016-10-26 (Estimated); Results first posted 2019-03-20 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-03

CONDITIONS: Head and Neck Neoplasms; Head and Neck Lymphedema; Head and Neck Cancer
Keywords: Lymphedema; Cancer; Head Cancer; Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Lymphedema; Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pneumatic Compression-1 session per day (Experimental): Head and neck garments for pneumatic compression device for treatment of lymphedema (1 session per day) with imaging using NIRFLI with ICG (Indocyanine green).
  Interventions: Device: Head and neck garments for pneumatic compression device; Drug: NIRFLI with ICG
- Pneumatic Compression-2 sessions per day (Experimental): Head and neck garments for pneumatic compression device for treatment of lymphedema (2 sessions per day) with imaging using NIRFLI with ICG (Indocyanine green).
  Interventions: Device: Head and neck garments for pneumatic compression device; Drug: NIRFLI with ICG

INTERVENTIONS:
Device: Head and neck garments for pneumatic compression device — Pneumatic compression device cleared for use by patients who are under medical supervision for the treatment of 1) lymphedema (primary or secondary); 2) edema resulting from mastectomies, trauma, sports injuries or post immobilization; 3) venous insufficiencies; 4) wounds; and 5) stasis dermatitis, venous stasis ulcers, arterial leg ulcers and diabetic foot ulcers and treatment of head and neck lymphedema
  Other Names: Flexitouch system
Drug: NIRFLI with ICG — Near-infrared Fluorescence Lymphatic Imaging following the off-label use of Indocyanine Green as a lymph contrast agent and the use of a custom designed fluorescence imager to dynamically follow lymphatic movement in subjects.
  Other Names: Near Infrared Fluorescence Imaging with Indocyanine Green

SUMMARY:
Assessment of lymphatic structure and function pre- and post- treatment and during recovery in head and neck cancer related lymphedema patients using NIR fluorescence lymphatic imaging: Response to ICD therapy in HNC Patients.

DETAILED DESCRIPTION:
A non-randomized, non-blinded, single site pilot study designed to assess whether near-infrared fluorescence imaging can report on the efficacy of a pneumatic compression device to move lymph in head and neck cancer survivors with resulting head and neck lymphedema.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years of age or older
* Participants must be diagnosed with Lymphedema of the Head and/or Neck
* Participants must be diagnosed with squamous cell carcinoma of the oral cavity, oropharynx or larynx and underwent surgery and radiation as part of their standard-of-care treatment plan.
* Participants must be ≥ 4 weeks post-radiation therapy
* Female participants of childbearing potential must have a negative urine pregnancy test ≤ 36 hours prior to study drug administration
* Female participants of childbearing potential must agree to use a medically accepted method of contraception for a period of one month after each imaging session
* Participants must be willing to use the Flexitouch® System at home daily for two (2) weeks

Exclusion Criteria:

* Women who are pregnant or breast-feeding
* Persons who are allergic to iodine
* A female of child-bearing potential, who does not agree to use an approved contraceptive for one month after study participation
* Persons who do not meet inclusion criteria
* Persons with pulmonary edema, thrombophlebitis, congestive heart failure, deep vein thrombosis, episodes of pulmonary embolism, infections and inflammation, or acute cancer
* Persons with uncontrolled hyperthyroidism or parathyroidism (for with an endocrinologist recommends against neck compression)
* Carotid sinus hypersensitivity syndrome
* Symptomatic carotid artery disease, as manifested by a recent transient ischemic attack (within 30 days), ischemic stroke, or amaurosis fugax (monocular visual ischemic symptoms or blindness)
* Symptomatic bradycardia in the absence of a pacemaker
* Internal jugular venous thrombosis, acute or within 3 months
* Known intracranial pressure or other contraindication to internal or external jugular venous compression
* Acute radiation dermatitis, unhealed surgical scar, unhealed or open wound(s), surgical flap less than 6-8 weeks post-operative
* Facial or head and neck dermal metastasis
* Acute facial infection (e.g., facial or parotid gland abscess)
* Any condition where increased venous and lymphatic return is undesirable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Rasmussen, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- UT Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Pneumatic Compression-1 Session Per Day: Head and neck garments for pneumatic compression device for treatment of lymphedema (1 session per day) with imaging using NIRFLI with ICG (Indocyanine green).
  Head and neck garments for pneumatic compression device.: Pneumatic compression device cleared for use by patients who are under medical supervision for the treatment of 1) lymphedema (primary or secondary); 2) edema resulting from mastectomies, trauma, sports injuries or post immobilization; 3) venous insufficiencies; 4) wounds and 5) stasis dermatitis, venous stasis ulcers, arterial leg ulcers and diabetic foot ulcers and treatment of head and neck lymphedema
  NIRFLI with ICG: Near-infrared Fluorescence Lymphatic Imaging following the off-label use of Indocyanine Green as a lymph contrast agent and the use of a custom designed fluorescence imager to dynamically follow lymphatic movement in subjects.
- Pneumatic Compression-2 Sessions Per Day: Head and neck garments for pneumatic compression device for treatment of lymphedema (2 sessions per day) with imaging using NIRFLI with ICG (Indocyanine green).
  Head and neck garments for pneumatic compression device.: Pneumatic compression device cleared for use by patients who are under medical supervision for the treatment of 1) lymphedema (primary or secondary); 2) edema resulting from mastectomies, trauma, sports injuries or post immobilization; 3) venous insufficiencies; 4) wounds and 5) stasis dermatitis, venous stasis ulcers, arterial leg ulcers and diabetic foot ulcers and treatment of head and neck lymphedema
  NIRFLI with ICG: Near-infrared Fluorescence Lymphatic Imaging following the off-label use of Indocyanine Green as a lymph contrast agent and the use of a custom designed fluorescence imager to dynamically follow lymphatic movement in subjects.
Period: Overall Study
Arm/Group | Pneumatic Compression-1 Session Per Day | Pneumatic Compression-2 Sessions Per Day
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pneumatic Compression-1 Session Per Day | Pneumatic Compression-2 Sessions Per Day | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 0 | 4
  >=65 years | 2 | 5 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 6 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 4 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Lymph Movement Measured by ICG Lymphography.
Description: Demonstrate the ability of the Flexitouch system to move lymph/enhance lymphatic uptake (indicated by increased functionality of vessels and/or changes in area of dermal backflow) as measured by Indocyanine Green (ICG) lymphography.
Time Frame: Single Treatment, 2 Weeks of Treatment
Population: The analysis population included all enrolled subjects who completed the study and properly used the device. One subject reported wearing the head garment upside down during the two week treatment period, therefore the subject was excluded from the analysis population for a cohort of 10 analyzable data sets.
Measure: Count of Participants; unit: Participants
Arm/Group | Pneumatic Compression-1 Session Per Day | Pneumatic Compression-2 Sessions Per Day
Number analyzed (Participants) | 5 | 5
Participants
  Lymph Movement after Single Treatment: Enhanced Lymphatic Uptake | 5 | 5
  Lymph Movement after Single Treatment: No Enhanced Lymphatic Uptake | 0 | 0
  Lymph Movement after 2 Weeks of Treatment: Enhanced Lymphatic Uptake | 5 | 4
  Lymph Movement after 2 Weeks of Treatment: No Enhanced Lymphatic Uptake | 0 | 1

2. Secondary Outcome: Dermal Backflow Measured by ICG Lymphography.
Description: Resolves dermal backflow as measured by ICG lymphography. A positive change in area indicates an increase in observable abnormal lymphatics, while a negative change indicates a decrease in observable abnormal lymphatics. A positive increase after a single treatment is expected as the manual stimulation of the lymphatics promotes the movement of ICG through the lymphatic space; however, a decrease over time provides an indication of improved lymphatic recovery.
Time Frame: Single Treatment, 2 Weeks of Treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pneumatic Compression-1 Session Per Day | Pneumatic Compression-2 Sessions Per Day
Number analyzed (Participants) | 5 | 5
Participants
  Dermal Backflow after Single Treatment): Positive Change in Area | 4 | 4
  Dermal Backflow after Single Treatment): Negative Change in Area | 0 | 0
  Dermal Backflow after Single Treatment): No Dermal Backflow/No Change | 1 | 1
  Dermal Backflow after 2 Weeks of Treatments: Positive Change in Area | 1 | 1
  Dermal Backflow after 2 Weeks of Treatments: Negative Change in Area | 3 | 3
  Dermal Backflow after 2 Weeks of Treatments: No Dermal Backflow/No Change | 1 | 1

3. Secondary Outcome: Symptom Alleviation Measured by Survey Response.
Description: Alleviates lymphedema symptoms as measured by survey response.
Time Frame: Single Treatment, 2 Weeks of Treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pneumatic Compression-1 Session Per Day | Pneumatic Compression-2 Sessions Per Day
Number analyzed (Participants) | 5 | 5
Participants
  After Single Treatment: Felt much better | 0 | 2
  After Single Treatment: Felt somewhat better | 4 | 2
  After Single Treatment: Felt about the same | 1 | 1
  After Single Treatment: Data Missing | 0 | 0
  After 2 Weeks of Treatment: Felt much better | 0 | 0
  After 2 Weeks of Treatment: Felt somewhat better | 2 | 4
  After 2 Weeks of Treatment: Felt about the same | 3 | 0
  After 2 Weeks of Treatment: Data Missing | 0 | 1

4. Secondary Outcome: Ease of Use Measured by Survey Response.
Description: Flexitouch is easy to use as measured by survey responses.
Time Frame: Single Treatment, 2 Weeks of Treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pneumatic Compression-1 Session Per Day | Pneumatic Compression-2 Sessions Per Day
Number analyzed (Participants) | 5 | 5
Participants
  Ability to Don after Single Treatment: Independently | 1 | 1
  Ability to Don after Single Treatment: Minimal Assist | 4 | 4
  Ability to Don after Single Treatment: Data Missing | 0 | 0
  Ability to Don after 2 Weeks of Treatment: Independently | 4 | 4
  Ability to Don after 2 Weeks of Treatment: Minimal Assist | 1 | 0
  Ability to Don after 2 Weeks of Treatment: Data Missing | 0 | 1
  Ability to Doff after Single Treatment: Independently | 4 | 3
  Ability to Doff after Single Treatment: Minimal Assist | 1 | 1
  Ability to Doff after Single Treatment: Data Missing | 0 | 1
  Ability to Doff after 2 Weeks of Treatment: Independently | 4 | 3
  Ability to Doff after 2 Weeks of Treatment: Minimal Assist | 1 | 0
  Ability to Doff after 2 Weeks of Treatment: Data Missing | 0 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment through study exit which was equivalent to approximately two weeks.
Arm/Group | Pneumatic Compression-1 Session Per Day | Pneumatic Compression-2 Sessions Per Day
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 3/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pneumatic Compression-1 Session Per Day (N=6) | Pneumatic Compression-2 Sessions Per Day (N=5)
Pain/Discomfort (Nervous system disorders) | 0 (0) | 1 (1) — Skin irritation on day 11 of use.
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Erythema around 3 ICG injection sites.
Infection (fungal) (Infections and infestations) | 0 (0) | 1 (1) — Oral thrush.

LIMITATIONS AND CAVEATS:
One subject reported wearing the head garment upside down during the two week treatment period, therefore the subject was excluded from the analysis population and replaced with another subject to meet the requirement for 10 analyzable data sets.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-04): https://cdn.clinicaltrials.gov/large-docs/21/NCT02946021/Prot_SAP_000.pdf